CLINICAL TRIAL: NCT06613542
Title: Effect Of Daily Taurine Supplementation For 6 Months On Biological Age and Metabolic Biomarkers As Well As Physical Fitness In 55-75-year-old Women And Men: A Randomized Controlled Intervention Study
Brief Title: Effects Of Daily Taurine Intake For 6 Months On Biological Age and Body Metabolism Indicators As Well As Physical Fitness In 55-75-year-old Women And Men
Acronym: TauAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Stanford University (Other); Rutgers University (Other); Universitaet Innsbruck (Other); LMU Klinikum (Other)
Responsible Party: Principal Investigator, Karolina Alicja Starzynska, Prof. Dr. med. Hans Hauner, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-253-S-CB
Record Dates: First submitted 2024-09-17; First posted 2024-09-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Taurine; Aging, Biological; Physical Activity; Metabolic Health; Anti-Aging; Longevity; Dietary Supplement; DNA Methylation; Sport
Keywords: taurine; biological aging; metabolic health; anti-aging; epigenetic clock; aging; physical activity; cognition; Cellular Senescence; hallmarks of aging; humans; Dietary Supplements; longevity; Taurine Deficiency; Taurine Level; aging metabolism; longevity physiology; drug effects; DNA-methylation; aging ptoeomics; DNA methylation; taurine microbiome; taurine gut micorbiota; taurine cognition; taurine sport; taurine DNA methylation; nutritional medicine; sport biology; taurine physical fitness; taurine physical acitvity; taurine sport biology; taurine muscle strength; taurine pwc 130; Taurine HOMA IR; taurine mental health; taurine human aging; taurine cardiometabolic risk; taurine cardiometabolic health; taurine blood pressure; taurine fasting glucose; taurine inflammation; taurine biological aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4g of taurine daily (Active Comparator): Intervention group (4g of taurine/day):
  2g of taurine (4 capsules, 500mg each) in the morning and 2g of taurine (4 capsules, 500mg each) in the evening for 6 months
  Interventions: Dietary Supplement: 4g of taurine daily
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 4g of taurine daily — Intervention group (4g of taurine/day): 2g of taurine (4 capsules, 500mg each) in the morning and 2g of taurine (4 capsules, 500mg each) in the evening for 6 months
  Arms: 4g of taurine daily
Dietary Supplement: Placebo — Controll group (4g of placebo/day): 2g of placebo (4 capsules, 500mg each) in the morning and 2g of placebo (4 capsules, 500mg each) in the evening for 6 months
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effect of taking 4 grams of taurine by older adults on aging processes over a period of 6 months. It will also check for effects of taurine on participant's physical fitness, metabolic and cognitive functions. The main question it aims to answer is:

• Does a supplementation with 4 g of taurine daily over a period of 6 months slow down biological aging in humans? Researchers will compare supplementation with taurine to a placebo (a look-alike substance that contains no drug) to reliably determine whether taurine has an effect.

Participants will:

* Take 4g of taurine or a placebo every day for 6 months
* Visit the study site 4 times for checkups and tests: for a screening visit, at the beginning of the intervention, after 8 and 24 weeks

DETAILED DESCRIPTION:
Measurements performed during study visits:

* Biological age estimate via proteome analysis
* Organ age estimates (proteomics)
* DNA methylation
* Inflammatory biomarkers (CRP, cytokines)
* Metabolic variables: fasting blood glucose, insulin, HOMA-IR, HbA1c, lipids, BMI
* Physical fitness (hand grip strength, leg extensor strength, PWC130)
* Resting energy expenditure
* Cognitive function via questionnaire
* Quality of life
* Heart rate variability
* Physical activity, nutrition

ELIGIBILITY:
Inclusion Criteria:

* women or men
* Age 55 - 75
* BMI 22 - 30 kg/m²
* written consent

Exclusion Criteria:

* Acute or chronic inflammation (e.g. flu infection)
* Severe chronic illness (e.g., Type 1 or Type 2 diabetes mellitus, COPD, renal insufficiency)
* Myocardial infarction or stroke in the previous 6 months
* Psychiatric disorder, including depression or dementia
* Weight change of ≥ 5 kg in the last 6 months

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Biological Age At 6 Months (Proteome Analysis) | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  The primary objective of the study is to answer the following research question:
  Does a 6-month supplementation with 4g of taurine daily slow down biological aging in humans?
  Biological age will be determined using a plasma proteome analysis and established machine learning models based on plasma and urine samples. This will also include an analysis of organ-specific aging.
Change From Baseline in Biological Age At 6 Months (DNA Methylation) | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  The primary objective of the study is to answer the following research question:
  Does a 6-month supplementation with 4g of taurine daily slow down biological aging in humans?
  Biological age will be estimated by assessing DNA methylation patterns (epigenetic clock) from plasma, urine, and oral mucosa samples.

SECONDARY OUTCOMES:
Change From Baseline In Cognitive Functions at 6 Months | pre-intervention (at time point 0) and post-intervention (after 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily influence parameters of mental health?
  Methods of measurement: MoCA (Montreal Cognitive Assessment)
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: fasting blood glucose in mg/dL
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: Body-Mass-Index determined by participants weight in kilograms divided by height in metres squared.
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: blood pressure in mmHg
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: total cholesterol in mg/dl
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: LDL-cholesterol in mg/dL
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: HDL-cholesterol in mg/dL
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: C-reactive protein in mg/l
Change From Baseline In Cardiometabolic Risk Profile at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Does a 6-month supplementation with 4 g of taurine daily alter the cardiometabolic risk profile?
  Measurement: fasting insulin in pmol/l
Change From Baseline In Handgrip Strength (kg) at 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Measurement of handgrip strength in kilograms and Newtons in the dominant hand using Jamar Hydraulic Hand Dynamometer.
Change From Baseline In Physical Working Capacity (PWC130) At 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Measurement of heart rate (bpm) on the Corvial ergometer while increasing power manually by 25 W every 2 minutes. The endpoint is the power in Watts at the stage where heart rate of 130bpm is reached.
Change From Baseline In Isometric Leg Extensor Strength For Each Leg At 6 Months | pre-intervention (at time point 0) and post-intervention (at 24 weeks)
  Measurement of leg extensor strength using a force transducer connected to the back of a chair and an ankle loop, as well as force recording software. The maximum force (N) will be multiplied with the distance from knee joint to the middle of the loop (in metres) to calculate the torque in Newton-metres (Nm) for each leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Nutritional Medicine of Technical University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of data privacy and confidentiality.

REFERENCES:
- [Background] Oh HS, Rutledge J, Nachun D, Palovics R, Abiose O, Moran-Losada P, Channappa D, Urey DY, Kim K, Sung YJ, Wang L, Timsina J, Western D, Liu M, Kohlfeld P, Budde J, Wilson EN, Guen Y, Maurer TM, Haney M, Yang AC, He Z, Greicius MD, Andreasson KI, Sathyan S, Weiss EF, Milman S, Barzilai N, Cruchaga C, Wagner AD, Mormino E, Lehallier B, Henderson VW, Longo FM, Montgomery SB, Wyss-Coray T. Organ aging signatures in the plasma proteome track health and disease. Nature. 2023 Dec;624(7990):164-172. doi: 10.1038/s41586-023-06802-1. Epub 2023 Dec 6. PMID 38057571
- [Background] Singh P, Gollapalli K, Mangiola S, Schranner D, Yusuf MA, Chamoli M, Shi SL, Lopes Bastos B, Nair T, Riermeier A, Vayndorf EM, Wu JZ, Nilakhe A, Nguyen CQ, Muir M, Kiflezghi MG, Foulger A, Junker A, Devine J, Sharan K, Chinta SJ, Rajput S, Rane A, Baumert P, Schonfelder M, Iavarone F, di Lorenzo G, Kumari S, Gupta A, Sarkar R, Khyriem C, Chawla AS, Sharma A, Sarper N, Chattopadhyay N, Biswal BK, Settembre C, Nagarajan P, Targoff KL, Picard M, Gupta S, Velagapudi V, Papenfuss AT, Kaya A, Ferreira MG, Kennedy BK, Andersen JK, Lithgow GJ, Ali AM, Mukhopadhyay A, Palotie A, Kastenmuller G, Kaeberlein M, Wackerhage H, Pal B, Yadav VK. Taurine deficiency as a driver of aging. Science. 2023 Jun 9;380(6649):eabn9257. doi: 10.1126/science.abn9257. Epub 2023 Jun 9. PMID 37289866